CLINICAL TRIAL: NCT04055870
Title: Efficacy, Safety, and Adequacy of EUS-guided Liver Biopsy
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 045.GID.2017.D
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Chronic Hepatic; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undergone EUS-guided liver biopsy at MDMC: Undergone EUS-guided liver biopsy at MDMC
  Interventions: Procedure: EUS-guided liver biopsy at MDMC

INTERVENTIONS:
Procedure: EUS-guided liver biopsy at MDMC — Endoscopic ultrasound (EUS) guided liver biopsy sampling is emerging as an alternative to the aforementioned approaches that offers several advantages, including decreased sampling variability and procedure-related complications.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and adequacy of EUS-guided liver biopsy in patients undergoing EUS-guided liver biopsy at Methodist Dallas Medical Center (MDMC).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy, safety, and adequacy of EUS-guided liver biopsy in patients undergoing EUS-guided liver biopsy at Methodist Dallas Medical Center (MDMC). This is a clinical quality improvement (CQI) initiative to evaluate outcomes within our institution. The data collected will be used to inform new innovative ways to improve EUS-guided liver biopsy with an ultimate goal of improving the quality of patient care. The clinical outcomes of this patient population have not been previously systematically reviewed in MDMC. Currently, the procedure in not being performed routinely at Methodist Dallas Medical Center (MDMC). However, with new technical and physician expertise, this option is now available at our institution. PI will evaluate the efficacy, safety, and adequacy of EUS-guided liver biopsy in patients requiring histologic examination of their liver at MDMC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergone EUS-guided liver biopsy at MDMC

Exclusion Criteria:

* Below 18 years of age
* Did not undergo EUS-guided liver biopsy at MDMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 18 years or older and have undergone EUS-guided liver biopsy at MDMC
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Length of core biopsy | 9/1/2017 and 9/1/2019
Number of portal tracts | 9/1/2017 and 9/1/2019
Diagnostic yield | 9/1/2017 and 9/1/2019
  We will define an adequate specimen as one containing ≥11 portal tracts or measuring ≥20 mm cumulative core length.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States